CLINICAL TRIAL: NCT02615080
Title: A Double-Blind, Randomised, Placebo-controlled, Parallel Group, International, Multi-centre Phase 2 Trial Investigating the Safety and Efficacy of CRD007 in Adult Subjects With Asthma
Brief Title: Safety and Efficacy of CRD007 in Adult Asthma Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: RSPR Pharma AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RSPR-008
Record Dates: First submitted 2015-11-17; First posted 2015-11-25 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CRD007 (Active Comparator): CRD007 (containing pemirolast sodium) tablets given twice daily for 14 weeks
  Interventions: Drug: CRD007
- Placebo (Placebo Comparator): Matching placebo tablets given given twice daily for 14 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CRD007
  Other Names: Pemirolast sodium
  Arms: CRD007
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a double-blind, randomised, placebo-controlled, parallel group, Phase 2 trial evaluating CRD007 administered orally b.i.d for 14 weeks for the treatment of asthma. CRD007 will be given as add on to a background of commonly used controller medication, i.e. inhaled corticosteroid (ICS) with or without long-acting beta2-agonist (LABA). By gradually reducing the background controller medication, the efficacy and safety of CRD007 will be evaluated on top of several dose levels of this medication.

DETAILED DESCRIPTION:
The present trial will include subjects with diagnosed asthma. The trial involves a total of 11 visits (Visit 1-2 are screening visits, visit 3 randomisation visit, visits 4-10 treatment visits and visit 11 follow-up visit).

The subjects will be monitored by medically qualified staff every second week at clinic visits, where the reduction of their background controller medication will be reduced, if their asthma is controlled.

Between visits to the clinic the subjects have to complete a diary.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age ≥18 years old
* Diagnosis of asthma according to Global Initiative for Asthma (GINA) Guidelines
* Atopic phenotype as assessed by the investigator
* Treated with ICS and LABA for at least 12 weeks prior to Visit 1with protocol defined daily doses
* Blood eosinophils ≥0.15*109/L at Visit 1
* Demonstration of forced expiratory volume at one second (FEV1) >60% of the predicted value at Visit 1
* Demonstration of ACQ6 ≥ 0.5 and ≤1.5 at Visit 1
* Reversibility of at least 12% and 200 mL in FEV1

Exclusion Criteria:

* Lower respiratory tract infection <6 weeks prior to Visit 1
* Current smokers
* Significant concurrent, uncontrolled medical condition as defined by the protocol
* Others, as defined in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2015-11-30 (Actual); Primary Completion 2017-02-21 (Actual); Study Completion 2017-02-24 (Actual)

PRIMARY OUTCOMES:
Change in ICS dose | Change of average dose of ICS, measured at visit 5 (week 8) and Visit 10 (week 18)

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke Backer, MD, Principal Investigator — Bispebjerg Hospital
Locations (24):
- Bulgaria (7):
  - MHAT St. Ivan Rilski-2003 Ltd., Department of Internal Medicine, Dupnitsa
  - SHATPPD - Pazardzhik EOOD, Department of phthisiatrics pneumonia and pulmonary functional diagnostics, Pazardzhik
  - Medical Center - Razgrad OOD, Office of Pneumonology and Phthisiatry, Razgrad
  - Medical Center Smolyan OOD, Office of Clinical Allergology, Smolyan
  - First MHAT - Sofia EAD, Third Department of Internal Medicine, Sofia
  - MHAT Lyulin EAD, Department of Internal Medicine, Sofia
  - SHATPPD Vratsa Ltd, Department of Pneumology, Vratsa
- Denmark (5):
  - Aalborg Universitetshospital, Aalborg
  - Hvidovre Hospital, Hvidovre
  - Bisbebjerg Hospital, København NV
  - Næstved Sygehus, Lungemedinsk afdeling, Næstved
  - Regionshospitalet Silkeborg, Silkeborg
- Poland (8):
  - Centrum Badań Klinicznych PI-House Sp. Z O.O., Gdansk
  - Medica Pro Familia, Katowice
  - NZOZ Centrum Medcyczne ProMiMed, Krakow
  - Medica Pro Familia, Krákow
  - Clinical Best Solution, Lublin
  - NZOZ ALERGO-MED. Specjalistyczna Przychodnia Lekarska, Poznan
  - Medica Pro Familia, Warsaw
  - Centrum Medyczne Oporów, Wroclaw
- United Kingdom (4):
  - The Medicines Evaluation Unit (MEU) Ltd, Manchester
  - Medinova North London Clinical Studies Center, Northwood
  - Medinova East London Clinical Studies Centre, Romford
  - Medinova South London Clinical Studies Centre, Sidcup